CLINICAL TRIAL: NCT01846416
Title: A Phase II, Multicenter, Single-arm Study of MPDL3280A in Patients With PD-L1-Positive Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Participants With Programmed Death-Ligand 1 (PD-L1) Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) [FIR]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28625; 2013-000177-69 (EudraCT Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

ARMS (3):
- Atezolizumab (MPDL3280): 1L Participants (Experimental): Participants with no prior chemotherapy for advanced NSCLC disease will receive atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until disease progression.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody
- Atezolizumab (MPDL3280): 2L+ Participants (Experimental): Participants who progress during or following a prior platinum-based chemotherapy regimen without restriction to maximum number of prior therapies will receive atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody
- Atezolizumab (MPDL3280): 2L+ Brain Metastases Participants (Experimental): Participants with previously treated brain metastases and who progress during or following a prior platinum-based chemotherapy regimen without restriction to the maximum number of prior therapies, will receive atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody — Atezolizumab 1200 mg IV on Day 1 of each 21-day cycle until disease progression.

SUMMARY:
This multicenter, single-arm study will evaluate the efficacy and safety of atezolizumab (MPDL3280A) in participants with PD-L1-positive locally advanced or metastatic NSCLC. Participants will receive an intravenous (IV) dose of 1200 milligrams (mg) atezolizumab (MPDL3280A) on Day 1 of 21-day cycles until disease progression.

Eligible participants will be categorized in to three groups as follows:

1. Participants with no prior chemotherapy for advanced disease;
2. Participants who progress during or following a prior-platinum based chemotherapy regimen for advanced disease (2L+participants);
3. Participants who are 2L+ and previously treated for brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB (not eligible for definitive chemoradiotherapy), Stage IV, or recurrent NSCLC
* PDL1-positive status as determined by an immunohistochemistry assay performed by a central laboratory. A positive result in chemotherapy, chemoradiation of the tumor sample biopsy will satisfy the eligibility criterion
* Eastern Cooperative Oncology group Performance Status of 0 or 1
* Life expectancy greater than or equal to 12 weeks
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors Version 1.1
* Adequate hematologic and end organ function

Exclusion Criteria:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment; the following exceptions are allowed. Hormone-replacement therapy or oral contraceptives, and tyrosine kinase inhibitors approved for treatment of NSCLC discontinued greater than 7 days prior to Cycle 1 Day 1
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Known central nervous system disease, including treated brain metastases in the following participants:

  1. who will not receive prior chemotherapy for advanced disease
  2. who progress during or following a prior-platinum based chemotherapy regimen for advanced disease (referred as 2L+ participants)
* Participants with a history of treated asymptomatic brain metastases are allowed in the 2L+ participants and previously treated for brain metastases.
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (31):
- United States (25):
  - HonorHealth Research Institute - Pima Center, Scottsdale, Arizona
  - Stanford University/Lucile Packard Children's Hospital, Palo Alto, California
  - The Angeles Clinic and Research Institute, Santa Monica Office, Santa Monica, California
  - University Of Colorado, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Hospital Cancer Inst, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists., St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Northwest Georgia Oncology Centers P.C., Carrollton, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dartmouth Hitchcock Med Center; Norris Cotton Cancer Ctr, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health Systems, Durham, North Carolina
  - Carolina BioOncology Institute; Can Therapy & Res Ctr, Huntersville, North Carolina
  - Ohio State Uni Hospital, Columbus, Ohio
  - Oncology Hematology Care, Inc., Hamilton, Ohio
  - Penn State Univ. Milton S. Hershey Medical Center; MSHMC Cardiology, Hershey, Pennsylvania
  - Penn Presbyterian Medical Center; Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI-Tennessee Oncology, Nashville, Tennessee
  - Huntsman Cancer Institute; University of Utah, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- Sint Augustinus Wilrijk, Wilrijk, Belgium
- Centre Léon Bérard, Lyon, France
- Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- United Kingdom (3):
  - Queen Mary University of London, London
  - Royal Marsden Hospital - Fulham; Oncology Department, London
  - Royal Marsden Hospital - Fulham, London

REFERENCES:
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 201 participants were screened for clinical eligibility, out of which 63 participants were screen failures, and hence 138 participants were enrolled, and 137 participants received treatment.
Groups:
- Atezolizumab (MPDL3280) : 1L Participants: Participants with no prior chemotherapy for advanced NSCLC disease received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until disease progression.
- Atezolizumab (MPDL3280): 2L+ Participants: Participants who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to maximum number of prior therapies received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
- Atezolizumab (MPDL3280): 2L+ Brain Metastases Participants: Participants with previously treated brain metastases and who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to the maximum number of prior therapies, received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
Period: Treatment Phase
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280): 2L+ Participants | Atezolizumab (MPDL3280): 2L+ Brain Metastases Participants
Started | 31 | 93 | 13
Completed | 0 | 0 | 0
Not Completed | 31 | 93 | 13
Not completed — Death | 2 | 9 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 2
Not completed — Other | 1 | 5 | 1
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Adverse Event | 3 | 4 | 0
Not completed — Non-compliance | 0 | 2 | 0
Not completed — Study Terminated by Sponsor | 1 | 4 | 0
Not completed — Progressive Disease | 21 | 63 | 9
Period: Survival Follow-up
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280): 2L+ Participants | Atezolizumab (MPDL3280): 2L+ Brain Metastases Participants
Started | 28 | 80 | 12
Completed | 0 | 0 | 0
Not Completed | 28 | 80 | 12
Not completed — Death | 21 | 62 | 9
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 7 | 0
Not completed — Study Terminated by Sponsor | 2 | 8 | 0
Not completed — Other | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received any dose of atezolizumab during the study.
Groups:
- Atezolizumab (MPDL3280) : 2L+ Participants: Participants who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to maximum number of prior therapies received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
- Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants: Participants with previously treated brain metastases and who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to the maximum number of prior therapies, received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
- Total: Total of all reporting groups
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants | Total
Number analyzed (Participants) | 31 | 93 | 13 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.8) | 65.2 (9.3) | 63.8 (7.7) | 65.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 34 | 7 | 58
  Male | 14 | 59 | 6 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response According to Modified Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response was defined as a complete response (CR) or partial response (PR), as determined by investigator according to modified RECIST criteria. Modified RECIST was derived from RECIST v1.1 conventions and immune related response criteria. CR was defined as disappearance of all tumor lesions (target lesion [TL] and non-target lesion [non-TL]) and no new measurable or unmeasurable lesions, all lymph node short axes must be less than 10 millimeters (mm), and PR was defined as at least 30 percent (%) decrease in sum of diameter of TLs and all new measurable lesions since baseline in absence of CR, and both confirmed by consecutive assessment greater than or equal to 4 weeks from date first documented. Participants not meeting these criteria, including participants without at least one post-baseline response assessment were considered as non-responders.
Time Frame: Baseline, and Day 1 of Cycle 1 (21-day cycle), then every 6 weeks for the first 12 months and then every 9 weeks thereafter until disease progression (up to 20 months)
Population: Efficacy-evaluable population; all treated participants who received at least 1 dose of atezolizumab during study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants | 32 [17 to 51] | 21 [13 to 30] | 23 [5 to 54]

2. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 (v1.1)
Description: Objective response was defined as a CR or PR, as determined by the investigator according to RECIST v1.1. For TLs, CR was defined as disappearance of all TLs. Any pathological lymph nodes, whether target or non-target, must had reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameter of TLs, taking as reference the baseline sum of diameters, in absence of CR. For non-TLs, CR was defined as disappearance of all non-TLs and if applicable, normalization of tumor marker level. Participants not meeting these criteria, including participants without at least 1 post-baseline response assessment were considered as non-responders.
Time Frame: as for outcome 1
Population: Efficacy-evaluable population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants | 29 [14 to 48] | 19 [11 to 28] | 23 [5 to 54]

3. Secondary Outcome: Duration of Objective Response According to RECIST v1.1
Description: Duration of objective response was defined as time from initial occurrence of documented CR or PR until documented disease progression (using RECIST v1.1 as determined by investigator) or death, whichever occurred first. For TLs, CR was defined as disappearance of all TLs. Any pathological lymph nodes, whether target or non-target, must had reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in sum of diameter of TLs, taking as reference baseline sum of diameters, in absence of CR. Progressive disease was at least a 20% increase in sum of diameters of TLs, taking as reference smallest sum on study (nadir). For non-TLs, CR was defined as disappearance of all non-TLs and if applicable, normalization of tumor marker level. Progressive disease was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. Participants were censored at the date of last tumor assessment.
Time Frame: as for outcome 1
Population: Efficacy-evaluable population with a confirmed objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 9 | 17 | 3
months | 9.2 [2.3 to 30.4] | 17.0 [2.8 to 44.2] | NA [2.8 to 9.9] — Median DOR was not reached.

4. Secondary Outcome: Percentage of Participants With 6-Month Duration of Objective Response
Description: Duration of objective response at 6 months was defined as time from initial occurrence of documented CR or PR until Month 6. For TLs, CR was defined as disappearance of all TLs. Any pathological lymph nodes, whether target or non-target, must have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in sum of diameter of TLs, taking as reference baseline sum of diameters, in absence of CR. For non-TLs, CR was defined as disappearance of all non-TLs and if applicable, normalization of tumor marker level. Participants were censored at the date of last tumor assessment.
Time Frame: Month 6
Population: Efficacy-evaluable population with a confirmed objective response.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 8 | 15 | 3
percentage of participants | 75.0 | 91.7 | 66.7

5. Secondary Outcome: Percentage of Participants With Disease Progression or Death According to RECIST v1.1
Description: For TLs, progressive disease was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest sum on study (nadir). For non-TLs, progressive disease was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Baseline to the first occurrence of progression or death, whichever occurs earlier (up to 20 months)
Population: Efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants | 67.7 | 74.2 | 84.6

6. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST v1.1
Description: PFS was defined as time from randomization to first occurrence of documented disease progression (based on RECIST v1.1 criteria) or death due to any cause within 30 days of the last treatment, whichever occurs earlier as determined by investigator. For TLs, progressive disease was defined as at least a 20% increase in the sum of diameter of TLs, taking as reference the smallest sum on study (nadir). For non-TLs, progressive disease was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. In event of no disease progression or documented death, PFS was censored at date of last evaluable tumor assessment. Participants with no post-baseline tumor assessments were censored at the time of first dose plus 1 day.
Time Frame: Baseline to the first occurrence of progression or death, whichever occurs earlier (up to 20 months)
Population: Efficacy-evaluable population.
Measure: Median (Full Range); unit: months
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
months | 4.5 [0.9 to 37.9] | 2.7 [0.0 to 45.5] | 2.5 [1.0 to 11.3]

7. Secondary Outcome: Percentage of Participants With PFS at Month 6, Month 12 and Month 30 According to RECIST v1.1
Description: Percentage of participants who were progression free at Month 6 and 12 (based on RECIST v1.1) was reported. For TLs, progressive disease was defined as at least a 20% increase in the sum of diameter of TLs, taking as reference the smallest sum on study (nadir). For non-TLs, progressive disease was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Months 6, 12 and 30
Population: Efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants
  Month 6 | 33.50 | 32.29 | 15.38
  Month 12 | 20 | 23 | NA — Not estimable
  Month 30 | 13 | 10 | NA — Not estimable

8. Secondary Outcome: Percentage of Participants With Disease Progression or Death According to Modified RECIST
Description: For TLs, progressive disease was defined as at least a 20% increase in the sum of diameters of TLs and new measurable lesions, taking as reference the smallest sum recorded since treatment started.
Time Frame: Baseline to the first occurrence of progression or death, whichever occurs earlier (up to 20 months)
Population: Efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants | 58.1 | 66.7 | 69.2

9. Secondary Outcome: PFS According to Modified RECIST
Description: PFS according to modified RECIST was defined as time from first dose of atezolizumab to first occurrence of documented disease progression or death due to any cause, as determined by investigator for participants who discontinued at first documented radiographic progression. For participants who continued beyond first documented progression and had follow-up tumor assessment or death, PFS was defined as time from first dose of atezolizumab to subsequent radiographic progression or death. For TLs, progressive disease was defined as at least a 20% increase in the sum of diameters of TLs and new measurable lesions, taking as reference the smallest sum recorded since treatment started. In event of no disease progression or documented death, PFS was censored at date of last evaluable tumor assessment.
Time Frame: Baseline to the first occurrence of progression or death, whichever occurs earlier (up to 20 months)
Population: Efficacy-evaluable population.
Measure: Median (Full Range); unit: months
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
months | 5.5 [0.9 to 37.9] | 3.7 [0.0 to 45.5] | 4.3 [1.1 to 16.2]

10. Secondary Outcome: Percentage of Participants With PFS at Month 6, Month 12 and Month 30 According to Modified RECIST
Description: Percentage of participants who were progression free at Months 6 and 12 (according to modified RECIST). For TLs, progressive disease was defined as at least a 20% increase in the sum of diameters of TLs and new measurable lesions, taking as reference the smallest sum recorded since treatment started.
Time Frame: Months 6, 12 and 30
Population: Efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants
  Month 6 | 43.12 | 39.10 | 44.87
  Month 12 | 31 | 29 | 24
  Month 30 | 12 | 10 | NA — Not estimable

11. Secondary Outcome: Percentage of Participants With Death
Description: Participants were followed for survival throughout the study.
Time Frame: Baseline till death or up to 20 months, whichever occurred first
Population: Efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
percentage of participants | 74.2 | 76.3 | 76.9

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of the study drug to the time of death from any cause of the study. Participants who were still alive at the time of analysis were censored at the time of their last study assessment (for active participants) or at the last date known alive (for participants in follow-up). If no post-baseline data were available, OS was censored at the date of first treatment plus 1 day.
Time Frame: Baseline till death or up to 20 months, whichever occurred first
Population: Efficacy-evaluable population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab (MPDL3280) : 1L Participants | Atezolizumab (MPDL3280) : 2L+ Participants | Atezolizumab (MPDL3280) : 2L+ Brain Metastases Participants
Number analyzed (Participants) | 31 | 93 | 13
months | 14.4 [12.8 to 22.1] | 9.3 [5.8 to 17.6] | 6.8 [3.2 to 19.5]

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Atezolizumab
Time Frame: Pre-dose (0 hour) and 30 minutes after infusion on Day 1 of Cycle 1
Population: Pharmacokinetic- evaluable population: All treated participants with pharmacokinetic data at specified time points. Here, Number of participants analyzed = number of participants with available data for this outcome. Per planned analysis, pharmacokinetic data were not analyzed separately for each cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Atezolizumab (MPDL3280) : All Arms: All participants included in the study were reported.
Arm/Group | Atezolizumab (MPDL3280) : All Arms
Number analyzed (Participants) | 135
micrograms per milliliter (mcg/mL) | 405 (31.7)

14. Secondary Outcome: Minimum Plasma Concentration (Cmin) for Atezolizumab
Time Frame: Pre-dose (0 hour) on Day 1 of Cycles 2, 3, 4, 8, and 16
Population: Pharmacokinetic- evaluable population. Here, Number of participants analyzed = number of participants with available data for this outcome, and n= number of participants with available data at the specified time point. Per planned analysis, pharmacokinetic data were not analyzed separately for each cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Atezolizumab (MPDL3280) : All Arms
Number analyzed (Participants) | 125
mcg/mL
  Pre-dose Cycle 2 (Day 1) (n= 125) | 68.8 (55.3)
  Pre-dose Cycle 3 (Day 1) (n= 100) | 90.6 (136.6)
  Pre-dose Cycle 4 (Day 1) (n= 92) | 123 (136.9)
  Pre-dose Cycle 8 (Day 1) (n= 51) | 206 (45.9)
  Pre-dose Cycle 16 (Day 1) (n= 1) | 135 (NA) — Geometric co-efficient of variation was not calculated as only 1 participant was analyzed at the specified time point.

ADVERSE EVENTS:
Time Frame: Baseline until 20 months.
Description: All participants who received at least one dose of atezolizumab were included in analysis.
Groups:
- Atezolizumab (MPDL3280A) : 1L Participants: Participants with no prior chemotherapy for advanced NSCLC disease received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until disease progression.
- Atezolizumab (MPDL3280A) : 2L+ Participants: Participants who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to maximum number of prior therapies received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
- Atezolizumab (MPDL3280A) : 2L+ Brain Metastases Participants: Participants with previously treated brain metastases and who had progressed during or following a prior platinum-based chemotherapy regimen without restriction to the maximum number of prior therapies, received atezolizumab IV as a fixed dose of 1200-mg on Day 1 of each 21-day cycle until no longer deemed to be experiencing clinical benefit as assessed by the investigator.
Arm/Group | Atezolizumab (MPDL3280A) : 1L Participants | Atezolizumab (MPDL3280A) : 2L+ Participants | Atezolizumab (MPDL3280A) : 2L+ Brain Metastases Participants
Serious Adverse Events (participants affected / at risk) | 17/31 | 46/93 | 6/13
Other Adverse Events (participants affected / at risk) | 31/31 | 88/93 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (MPDL3280A) : 1L Participants (N=31) | Atezolizumab (MPDL3280A) : 2L+ Participants (N=93) | Atezolizumab (MPDL3280A) : 2L+ Brain Metastases Participants (N=13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 8 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 2
Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Thyroiditis acute (Endocrine disorders) | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0
AUTOIMMUNE COLITIS (Gastrointestinal disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0 | 0
INFLUENZA B VIRUS TEST POSITIVE (Investigations) | 1 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (MPDL3280A) : 1L Participants (N=31) | Atezolizumab (MPDL3280A) : 2L+ Participants (N=93) | Atezolizumab (MPDL3280A) : 2L+ Brain Metastases Participants (N=13)
Fatigue (General disorders) | 16 | 38 | 5
Pyrexia (General disorders) | 7 | 21 | 1
Oedema peripheral (General disorders) | 3 | 14 | 2
Chest pain (General disorders) | 1 | 9 | 0
Pain (General disorders) | 3 | 2 | 2
Asthenia (General disorders) | 1 | 9 | 0
Chills (General disorders) | 1 | 5 | 1
Influenza like illness (General disorders) | 3 | 4 | 1
Malaise (General disorders) | 0 | 6 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 27 | 4
Constipation (Gastrointestinal disorders) | 8 | 16 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 17 | 4
Vomiting (Gastrointestinal disorders) | 4 | 14 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 8 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5 | 1
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 33 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 30 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 18 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 19 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 8 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 9 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 22 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 12 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 12 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 7 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 8 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 6 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 12 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 9 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 17 | 0
Pneumonia (Infections and infestations) | 1 | 8 | 0
Urinary tract infection (Infections and infestations) | 7 | 3 | 2
Candida infection (Infections and infestations) | 2 | 1 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 4 | 11 | 1
Anxiety (Psychiatric disorders) | 0 | 11 | 2
Depression (Psychiatric disorders) | 3 | 9 | 1
Confusional state (Psychiatric disorders) | 1 | 4 | 1
Hallucination (Psychiatric disorders) | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 19 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 10 | 3
Dizziness (Nervous system disorders) | 4 | 8 | 1
Dysgeusia (Nervous system disorders) | 4 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Weight decreased (Investigations) | 6 | 9 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 2
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 9 | 0
Hypertension (Vascular disorders) | 3 | 3 | 1
Hot flush (Vascular disorders) | 0 | 2 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 1
Aortic valve thickening (Cardiac disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 2 | 1
Lacrimation increased (Eye disorders) | 0 | 2 | 1
Vision blurred (Eye disorders) | 2 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1
EXCESSIVE CERUMEN PRODUCTION (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 3 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 6 | 0
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 1 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 3 | 1
STOMATITIS (Gastrointestinal disorders) | 2 | 3 | 0
SINUSITIS (Infections and infestations) | 2 | 2 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
PARAESTHESIA (Nervous system disorders) | 2 | 4 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.